CLINICAL TRIAL: NCT07251595
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase II Clinical Study to Evaluate the Efficacy and Safety of SHR0302 Tablets as Single Therapy or in Combination With SHR0302 Base Gel in the Treatment of Patients With Non-segmental Vitiligo
Brief Title: A Trial of SHR0302 Tablets and SHR0302 Base Gel in Patients With Non-segmental Vitiligo
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR0302-202
Record Dates: First submitted 2025-11-19; First posted 2025-11-26 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Non-segmental Vitiligo
MeSH Terms: interventions — ivarmacitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- SHR0302 tablets in low dose group (Experimental)
  Interventions: Drug: SHR0302 Tablets; Drug: SHR0302 Base Placebo Gel
- SHR0302 tablets in high dose group (Experimental)
  Interventions: Drug: SHR0302 Tablets; Drug: SHR0302 Base Placebo Gel
- SHR0302 tablets + SHR0302 Base gel group (Experimental)
  Interventions: Drug: SHR0302 Tablets; Drug: SHR0302 Base Gel
- SHR0302 placebo tablets + SHR0302 Base placebo gel group (Placebo Comparator)
  Interventions: Drug: SHR0302 Placebo Tablets; Drug: SHR0302 Base Placebo Gel

INTERVENTIONS:
Drug: SHR0302 Tablets — SHR0302 tablets.
  Arms: SHR0302 tablets + SHR0302 Base gel group; SHR0302 tablets in high dose group; SHR0302 tablets in low dose group
Drug: SHR0302 Base Gel — SHR0302 Base gel.
  Arms: SHR0302 tablets + SHR0302 Base gel group
Drug: SHR0302 Placebo Tablets — SHR0302 placebo tablets.
  Arms: SHR0302 placebo tablets + SHR0302 Base placebo gel group
Drug: SHR0302 Base Placebo Gel — SHR0302 Base placebo gel.
  Arms: SHR0302 placebo tablets + SHR0302 Base placebo gel group; SHR0302 tablets in high dose group; SHR0302 tablets in low dose group

SUMMARY:
The study is being conducted to evaluate the efficacy, and safety of SHR0302 tablets as single therapy or in combination with SHR0302 Base gel for patients with non-segmental vitiligo.

ELIGIBILITY:
Inclusion Criteria:

1. Sign the informed consent form before the clinical trial.
2. On the day of signing the informed consent form, the age must be between 18 and 75 years old (inclusive), and it can be either male or female.
3. The subjects and their partners had no intention of having children during the study period and within one month after the administration of the drug, did not donate sperm or eggs, and voluntarily adopted effective contraceptive measures. The serum pregnancy test results of the female subjects must be negative and they must not be in the lactation period.
4. During the screening process, it was clinically diagnosed as non-segmental vitiligo.
5. Throughout the entire research process, the participants agreed to stop using all treatments related to vitiligo as well as any cosmetic products with therapeutic effects.

Exclusion Criteria:

1. Subjects diagnosed with segmental, mixed or undifferentiated vitiligo; or subjects previously diagnosed with other skin pigmentation disorders.
2. When the facial skin lesions caused by vitiligo cover more than 33% of the area with white hair.
3. During the screening period or at the baseline, there were other active skin lesions or skin infections that might interfere with the use of the study drug or the evaluation of the drug's efficacy.
4. Subjects with a history of related infections/communicable diseases or infection/contagion history.
5. Known or suspected history of immunosuppression.
6. Tuberculosis (TB) or latent tuberculosis infection.
7. Positive for human immunodeficiency virus antibody HIV-Ab, positive for syphilis-specific antibody, positive for hepatitis C virus antibody HCV-Ab, or hepatitis B virus (HBV) infection.
8. Subjects who have malignant tumors or have a history of malignant tumors.
9. Abnormal thyroid function, with a history of thrombotic diseases within the previous 12 months, and having experienced a cardiovascular or cerebrovascular event that required hospitalization within the previous 12 months.
10. There are serious abnormalities in the cardiovascular, mental, renal, liver, immune, gastrointestinal, urogenital, nervous, skeletal-muscular, skin, sensory, endocrine or hematological systems.
11. Pregnant women, lactating women, or female participants who plan to become pregnant during the study period.
12. Those who are known to be allergic to the test drug or any component of the test drug.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2025-12-05 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
The percentage change in the facial vitiligo area score index (F-VASI) from the baseline. | At Week 24.

SECONDARY OUTCOMES:
The percentage change in F-VASI compared to the baseline. | Up to 48 weeks.
  Except for Week 24.
The percentage change in the total body vitiligo area score index (T-VASI) compared to the baseline. | Up to 48 weeks.
The proportion of subjects who achieved an improvement of at least 50%/75%/90% compared to the baseline on the F-VASI (F-VASI 50/75/90 response). | Up to 48 weeks.
The proportion of subjects who achieved at least a 50%/75%/90% improvement in T-VASI compared to the baseline (T-VASI 50/75/90 response). | Up to 48 weeks.
The absolute change in facial vitiligo area (F-BSA) compared to the baseline. | Up to 48 weeks.
The percentage change in facial vitiligo area (F-BSA) compared to the baseline. | Up to 48 weeks.
The percentage change the total body vitiligo area (T-BSA) compared to the baseline. | Up to 48 weeks.
The absolute change the total body vitiligo area (T-BSA) compared to the baseline. | Up to 48 weeks.
The proportion of subjects who achieved a significant improvement (4) on the Vitiligo Visual Scale (VNS). | Up to 48 weeks.
The proportion of subjects who achieved a complete improvement (5) on the Vitiligo Visual Scale (VNS). | Up to 48 weeks.
The absolute values of the changes in the vitiligo-specific quality of life scale (VitiQoL) compared to the baseline. | Up to 48 weeks.
The percentages of the changes in the vitiligo-specific quality of life scale (VitiQoL) compared to the baseline. | Up to 48 weeks.
The proportion of subjects who achieved the facial - vitiligo physician global assessment (F-PhGVA) of no depigmentation (0). | Up to 48 weeks.
The proportion of subjects who achieved the facial - vitiligo physician global assessment (F-PhGVA) of almost no depigmentation (1). | Up to 48 weeks.
The proportion of subjects who achieved the overall assessment of vitiligo by dermatologists (T-PhGVA) as no depigmentation (0). | Up to 48 weeks.
The proportion of subjects who achieved the overall assessment of vitiligo by dermatologists (T-PhGVA) as almost no depigmentation (1). | Up to 48 weeks.
The proportion of subjects who achieved a significant improvement (1) in the facial vitiligo condition as perceived by the overall impression (F-PaGIC-V). | Up to 48 weeks.
The proportion of subjects who achieved a moderate improvement (2) in the facial vitiligo condition as perceived by the overall impression (F-PaGIC-V). | Up to 48 weeks.
The proportion of subjects who achieved a significant improvement (1) in the overall impression (T-PaGIC-V) of generalized vitiligo. | Up to 48 weeks.
The proportion of subjects who achieved a moderate improvement (2) in the overall impression (T-PaGIC-V) of generalized vitiligo. | Up to 48 weeks.
The plasma concentration of SHR0302. | Week 12 and Week 24.
The relative change in serum CXCL-9 level before administration compared to the baseline value. | At Week 4, 12, 24, 32, and 48.
The relative change in serum CXCL-10 level before administration compared to the baseline value. | At Week 4, 12, 24, 32, and 48.

CONTACTS AND LOCATIONS:
Locations (1):
- Dermatology Hospital affiliated to Shandong First Medical University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided